CLINICAL TRIAL: NCT04996849
Title: Contemporary Characteristics of Penile Carcinoma: at M.D. Anderson Cancer Center, and Harris Health System and Katy, Sugar Land, the Woodlands and Bay Area Regional Care Centers
Brief Title: Contemporary Characteristics of Penile Cancer
Status: Terminated | Type: Observational
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PCR04-0148; NCI-2021-07693 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PCR04-0148 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Penile Carcinoma; Squamous Cell Carcinoma of the Penis
MeSH Terms: conditions — Penile Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational (data collection): Patients undergo data collection every 6 months for up to 15 years.
  Interventions: Other: Data Capture; Other: Questionnaire Administration

INTERVENTIONS:
Other: Data Capture — Data collected
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This study develops a prospective database of patients who are evaluated and treated for penile cancer. This will facilitate analyzing trends in cancer incidence, risk factors, treatment, complications, and tumor progression. It will also prospectively validate the importance of pathological prognostic factors previously reported and outcome related to contemporary treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To prospectively collect data on the presenting features, management and outcome of penile carcinoma at M.D. Anderson Cancer Center, and Harris Health System and Katy, Sugar Land, The Woodlands and Bay Area Regional Care Centers.

OUTLINE:

Patients undergo data collection every 6 months for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* All diagnosed patients with a primary penile malignancy, including those with squamous carcinoma

Exclusion Criteria:

* No patient meeting the above criteria will be excluded

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with a primary penile malignancy
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2004-04-22 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Prospectively collect data on the presenting features, management and outcome of penile carcinoma | Up to 15 years
  Descriptive statistics will be utilized where applicable to address questions relevant to the study aims.

CONTACTS AND LOCATIONS:
Overall Officials: Curtis A Pettaway, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT04996849/ICF_000.pdf